CLINICAL TRIAL: NCT02074527
Title: Phase 0 _ Brazilian Registry of Congenital HeArt Disease INtervention and Angiography
Brief Title: CHAIN_brazilian Registry of Congenital HeArt Disease INtervention and Angiography
Acronym: CHAIN
Status: Completed | Type: Observational
Sponsor: Hospital do Coracao (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Other Study IDs: CAAE_08691912.8.1001.0060
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2014-02

CONDITIONS: Congenital Heart Disease; Cardiac Catheterization; Brazilian Electronic Registration; Catheterization Diagnostic or Therapeutic
Keywords: congenital heart disease; cardiac catheterization; brazilian electronic registration
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Design: Observational - Cross study with followed up for 30 days. The Primary Objective is to realize a record that reflects a national overview of the role of cardiac catheterization in patients with congenital heart disease in hospitals distributed by geographic density of each region of Brazil.

DETAILED DESCRIPTION:
Patients admitted in the hemodynamic sector with diagnosed or suspected congenital cardiopathy and undergoing diagnostic or therapeutic cardiac catheterization. Participants release the data in (e-CRF) electronics system. Sample: 2000 records.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hemodynamic sector with diagnosed or suspected congenital cardiopathy and undergoing diagnostic or therapeutic cardiac catheterization.

Exclusion Criteria:

* Patients undergoing hybrid approach to intervention, with the aid of cardiac surgery to realization of cardiac catheterization.

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the hemodynamic sector with diagnosed or suspected congenital cardiopathy and undergoing diagnostic or therapeutic cardiac catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of serious complications of cardiac catheterization in congenital heart | December 2014
  Occurrence of serious complications of cardiac catheterization in congenital heart procedure-related (occurring within 7 days after the procedure or until hospital discharge, whichever occurs first, and following 30 days), such as embolization of the prosthesis, cardiac arrhythmias, trauma vascular intracardiac injury, death, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Otavio Berwanger, São Paulo, Brazil